CLINICAL TRIAL: NCT02344264
Title: Effect of Nervus Cutaneous Femoris Lateralis-Blockade on Moderate Pain Responders After Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Hägi-Pedersen (Other)
Responsible Party: Sponsor-Investigator, Daniel Hägi-Pedersen, Consultant, Naestved Hospital
Organization: Naestved Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROTOKOL - 001-2014 - KHTY; 2014-003730-10 (EudraCT Number)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Pain, Postoperative; Ropivacaine; Therapeutic Use; Arthroplasty, Replacement, Hip
Keywords: US guided nerve block; Total hip Arthroplasty; NCFL; nervus cutaneous femoralis lateralis
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RP (Other): first blockade: ropivacaine 7,5mg/ml 8 ml second blockade: placebo: saline 8 ml
  Interventions: Drug: Ropivacaine; Drug: Saline
- PR (Other): first blockade: placebo: saline 8 ml second blockade: ropivacaine 7,5mg/ml 8 ml
  Interventions: Drug: Ropivacaine; Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Arm RP is receiving 8 ml of ropivacaine 7,5 mg/ml at first blockade (NCFL) and after 45 minutes another blockade (NCFL) with placebo (saline 8ml).
  Arm PR is receiving 8 ml of placebo (saline) at first blockade (NCFL) and after 45 minutes another blockade (NCFL) with ropivacaine 8 ml.
  Other Names: Naropin
Drug: Saline — Arm RP is receiving 8 ml of ropivacaine 7,5 mg/ml at first blockade (NCFL) and after 45 minutes another blockade (NCFL) with placebo (saline 8ml).
  Arm PR is receiving 8 ml of placebo (saline) at first blockade (NCFL) and after 45 minutes another blockade (NCFL) with ropivacaine 8 ml.
  Other Names: NaCl; Placebo

SUMMARY:
The patients will be included the 1. or 2. day after surgery. All THA patients will be screened. Those reporting VAS > 40 during active 30 degrees hip flexion will be asked to participate.

Included patients will receive 2xNCFL (singleshot) first placebo (8 ml saline) and then ropivacaine (8 ml ropivacaine 7,5mg/ml) or the other way around (randomized). There will be 45 minutes between the two blockades. The blockades will be ultrasound guided.

ELIGIBILITY:
Inclusion Criteria:

* THA within 48 hours and VAS>40 during active 30 degrees hip flexion despite conventional pain medication.
* informed consent
* ASA 1-3
* BMI 18-40

Exclusion Criteria:

* Unable to communicate in danish
* Allergic reactions toward drugs used
* Abuse of alcohol/drugs
* Unable to cooperate
* Pregnant women

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference in VAS between NCFL and placebo during active 30 degrees hip flexion | 45 min

SECONDARY OUTCOMES:
Difference in mean VAS between the groups during active hip flexion | 15, 30, 45, 60, 75, 90 min
Difference in mean VAS between the groups at rest | 15, 30, 45, 60, 75, 90 min

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hägi-Pedersen, Ph.D., Study Chair — Naestved Hospital, Department of Anaesthesiology
Locations (1):
- Department of Anaesthesiology, Næstved, Danmark, Denmark